CLINICAL TRIAL: NCT00520104
Title: A Randomized, Open Label, Single Center, Single-Dose Study to Assess the Effects of Certain Nasal Medications on the Pharmacokinetics, Safety and Tolerability of PMI-150 (Intranasal Ketamine Hydrochloride) 30 mg
Brief Title: Determination of Drug Interactions of Certain Nasal Medications With Intranasal Ketamine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KET-PK-008
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2007-08

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): intranasal ketamine
  Interventions: Drug: intranasal ketamine
- B (Experimental): oxymetazoline plus intranasal ketamine
  Interventions: Drug: intranasal ketamine
- C (Experimental): intranasal steroid plus intranasal ketamine
  Interventions: Drug: intranasal ketamine

INTERVENTIONS:
Drug: intranasal ketamine — drug interaction

SUMMARY:
This is an open label, single-center study to determine whether certain nasal medication interact with PMI-150 (intranasal ketamine) 30 mg in healthy adult volunteers and in patients with allergic rhinitis.

DETAILED DESCRIPTION:
To assess separately the effects of a nasal vasoconstrictor (oxymetazoline) and of a nasal steroid on the rate and extent of intranasal absorption of PMI-150 30 mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Patients with Allergic Rhinitis

Exclusion Criteria:

* Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics | multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (1):
- Javelin Pharmaceuticals, Cambridge, Massachusetts, United States